CLINICAL TRIAL: NCT06834971
Title: Colistin Methanesulfonate Sodium Inhalation for Prophylaxis of Ventilator-Associated Pneumonia (CIVAP): A Prospective, Multicentre, Double-Blind, Randomized, Placebo-Controlled Trial
Acronym: CIVAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wang Hao, professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Qilu Wang Hao
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Ventilator-Associated Pneumonia (VAP)
Keywords: colistin; prevention; nebulization
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMS group (Experimental): Participants were randomly assigned to receive either CMS (75mg caculated as colistin base activity(CBA), solubilized in 4 mL 0.9% saline) twice daily. Nebulization will be performed using a vibrating mesh nebulizer (Aeroneb solo, Aerogen, Galway, Ireland) placed in the inspiratory limb of the ventilator tubing, behind the Y-piece, and continued until the nebulizer deposit becomes dry for three consecutive days of mechanical ventilation. To ensure the experiment is conducted under blind conditions, the Nebulizer will be covered with an opaque protective cover. A filter will be placed on the expiratory limb to protect the ventilator.
  Interventions: Drug: Colistimethate sodium (CMS)
- NS group (No Intervention): Participants were randomly assigned to receive equivalent volume of 0.9% saline (NS group), twice daily. Nebulization will be performed using a vibrating mesh nebulizer (Aeroneb solo, Aerogen, Galway, Ireland) placed in the inspiratory limb of the ventilator tubing, behind the Y-piece, and continued until the nebulizer deposit becomes dry for three consecutive days of mechanical ventilation. To ensure the experiment is conducted under blind conditions, the Nebulizer will be covered with an opaque protective cover. A filter will be placed on the expiratory limb to protect the ventilator.

INTERVENTIONS:
Drug: Colistimethate sodium (CMS) — CMS (colistimethate sodium, 75mg, solubilized in 4 mL 0.9% saline), twice daily. Nebulization will be performed using a vibrating mesh nebulizer (Aeroneb solo, Aerogen, Galway, Ireland) placed in the inspiratory limb of the ventilator tubing, behind the Y-piece, and continued until the nebulizer deposit becomes dry for three consecutive days of mechanical ventilation. To ensure the experiment is conducted under blind conditions, the Nebulizer will be covered by stickers. A filter will be placed on the expiratory limb to protect the ventilator.
  Arms: CMS group

SUMMARY:
Previous studies have identified Acinetobacter baumannii (AB), Pseudomonas aeruginosa (PA), and Klebsiella pneumoniae (KP) as the predominant pathogens responsible for ventilator-associated pneumonia (VAP). The challenge of drug resistance, especially against carbapenem is intensifying, with variations noted across different regions. Multidrug-resistant organisms associated VAP (MDR-VAP) are increasing in frequency and are associated with significant morbidity, mortality, therefore imposes a heavy burden on the healthcare system. Colistin methanesulfonate sodium (CMS) has shown effectiveness against gram-negative bacteria, including carbapenem-resistant organisms (CRO) such as carbapenem-resistant Acinetobacter baumannii (CRAB), carbapenem-resistant Pseudomonas aeruginosa (CRPA), and carbapenem-resistant Klebsiella pneumoniae (CRKP). This trial aims to evaluate the efficacy of a 3-day course of inhaled CMS in lowering the incidence of VAP among patients undergoing invasive mechanical ventilation for at least two days and at high risk of MDR-VAP.

DETAILED DESCRIPTION:
Ventilator-Associated Pneumonia (VAP) is defined as pneumonia that develops 48-72 hours or more following the initiation of mechanical ventilation. It is a critical infection acquired in the Intensive Care Unit (ICU), significantly contributing to increased mortality rates, extended ICU stays, and elevated healthcare costs for patients on ventilators[1]. VAP is reported to affect 5-40% of patients receiving mechanical ventilation, with an average incidence of 20-25%. This proportion has been exacerbated in recent years by the COVID-19 pandemic[2-4]. A meta-analysis encompassing 195 studies found that the overall cumulative incidence of VAP in mainland China is 23.8% (95% CI 20.6-27.2%)[5].

Numerous risk factors, such as prolonged mechanical ventilation, advanced age, supine body position, prior antibiotic use, and various comorbidities, in addition to the endotracheal intubation itself, have been associated with the development of VAP[6, 7]. VAP results from the invasion of pulmonary parenchyma by pathogenic bacteria, which overwhelm the host's weakened defense capability. The primary sources of these bacteria include oropharyngeal colonization, secretions around the endotracheal tube cuff, and biofilm formation on the tracheal tube. The infectious process initiates at the time of intubation and progresses over several days. Reports indicate that the daily risk of VAP peaks between days 5 and 9 of incubation, underscoring the need for early preventive measures[8]. Despite decades of research highlighting interventions such as patient positioning adjustments, daily awakening and weaning protocols, oral decontamination, and systemic antibiotics to reduce VAP incidence, the burden remains unacceptably high.

Systemic antibiotics are commonly used for both treatment and prevention of VAP. However, the risk of resistant bacteria selection is a significant concern. A meta-analysis of six trials indicated that prophylactic antibiotics administered via nebulization effectively reduced VAP occurrence without increasing the risk of multidrug resistant (MDR) pathogen-related VAP[9]. Another Meta-Analysis consisting seven RCTs also confirmed that pro- phylactic antibiotics delivered via the respiratory tract reduced the risk of VAP, particularly for those treated with nebulized aminoglycosides[10]. Additionally, a short course of aerosolized ceftazidime significantly decreased VAP frequency in critically ill trauma patients without adversely affecting bacterial pathogen profiles and sensitivity patterns[11]. Recently, a study of 3-day course of inhaled amikacin was shown to effectively reduce the incidence of VAP[12, 13]. Stephan Ehrmann's team confirmed the possibility of inhaled amikacin to lessen the VAP burden during a 28-day follow-up period. This study provides us with excellent inspiration and suggests promising prospects for the use of nebulized antibiotics in preventing VAP. However, there are still more than 10% of patients who have amikacin resistance that can not be covered among all participants and the burden of MDR-VAP has becoming increasingly heavy with variations across different regions. Data from China Antimicrobial Surveillance Network (CHINET 2024) shows the resistance rates of Acinetobacter baumannii (AB), Klebsiella pneumoniae (KP), and Pseudomonas aeruginosa (PA) to amikacin are 49.5%, 15.5%, and 3.4%, respectively. In contrast, the resistance rates of carbapenem-resistant Acinetobacter baumannii (CRAB), carbapenem-resistant Klebsiella pneumoniae (CRKP), and carbapenem-resistant Pseudomonas aeruginosa (CRPA) to amikacin are as high as 77.4%, 67.1%, and 11.4%, respectively.

Given the effectiveness of CMS against gram-negative bacteria including carbapenem-resistant organisms (CRO), we are optimistic about the potential of nebulized CMS inhalation to prevent VAP. So we designed the study to evaluate the efficacy and safety of prophylactic CMS nebulization in preventing VAP among incubated patients at high risk of MDR-VAP. We hypothesize that administering a 3-day course of pre-emptive inhaled CMS after 2 days of ventilation will reduce the subsequent incidence of VAP.

ELIGIBILITY:
Participants will be enrolled if they meet the following criteria:

1. Age ≥18 years;
2. Mechanical ventilation for more than two consecutive days (48 hours);
3. Patient has high-risk factors for multidrug-resistant bacterial infections, which meet any of the following criteria:

(1)History of antibiotic exposure within 30 days; (2)Hospitalization time>5 days (120 hours); (3)Septic shock; (4) ARDS; (5)Accept renal replacement therapy; (6)Previous colonization of multidrug-resistant bacteria; 4. Informed consent of the patient or a proxy was written.

Participants will be excluded in case of:

1. Suspected or confirmed VAP at the inclusion day;
2. Patient ventilated through an endotracheal tube for more than four consecutive days (96 hours);
3. Expected that endotracheal intubation will be removed within the next 24 hours;
4. Tracheostomy;
5. Allergy to CMS;
6. Patients has polymyxins medication history within 7 days or clinical indication for systemic CMS therapy at the inclusion day;
7. Chronic kidney failure with baseline glomerular filtration ≤30 mL/min or Stage 3 classification AKI (KDIGO) (excluding patients undergoing renal replacement therapy);
8. Expected survival time not exceeding 48 hours;
9. Pregnancy or breastfeeding period;
10. Patients previously included in this study or are using any inhaled antibiotics or are participating in other clinical studies within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of a first VAP episode from randomization to day 28 | from randomization to day 28
  calculated as the ratio of the number of patients diagnosed VAP divided by the number of randomized patients in each group

SECONDARY OUTCOMES:
incidence of a first MDR-VAP episode from randomization to day 28 | from randomization to day 28
  Calculated as the ratio of the number of patients diagnosed VAP divided by the number of randomized patients in each group
Incidence density of adjudicated VAP from randomisation to day 28 | from randomization to day 28
  per 1000 patient-days of invasive mechanical ventilation
Incidence of gram-negative bacteria-related VAP with in vitro susceptibility to CMS from randomisation to day 28 | from randomization to day 28
  the incidence of ventilator-associated pneumonia due to gram-negative bacteria with in vitro susceptibility to colistin
The number of antibiotic-days from randomisation to day 28 | from randomization to day 28
  the sum of the number of systemic antibiotic treatments received each day
The number of days of mechanical ventilation from randomization to day 28 | from randomization to extubation or day 28, whichever occurs first
  the number of days of mechanical ventilation
The number of days in the ICU and hospital from randomization to day 90 | from randomization to day 90
  the number of days in the ICU and the hospital
Mortality at day 28 and 90 | from randomization to day 28 and day 90
  Mortality at 28- and 90-day after randomization
Evaluation of nebulization safety and side effects from randomisation to day 28 | from randomization to day 28
  Evaluation of nebulization safety and side effects: nephrotoxicity, neurotoxicity, and bronchospasm
Incidence of CMS-resistant bacteria in tracheobronchial aspirate (TBA) or blood from randomisation to day 28 | from randomization to day 28
  incidence of colistin-resistant bacteria in tracheobronchial aspirate (TBA) or blood
Incidence of ventilator-associated events from randomisation to extubation or day 28, whichever occurs first | from randomization to extubation or day 28, whichever occurs first
  Incidence of ventilator-associated events， including ventilator-associated conditions (VACs), infection-related ventilator associated complications (IVACs), and possible VAP (PVAP).

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Professor, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form will be shared with other researchers when start this trial.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and ICF will be shared with other researchers when start this trial for five years.
Access Criteria: Ever researchers can access our study protocol and ICF from the web of clinical trials.gov.

REFERENCES:
- [Background] Wu Z, Zhang S, Cao Y, Wang Q, Sun K, Zheng X. Comparison of the clinical efficacy and toxicity of nebulized polymyxin monotherapy and combined intravenous and nebulized polymyxin for the treatment of ventilator-associated pneumonia caused by carbapenem-resistant gram-negative bacteria: a retrospective cohort study. Front Pharmacol. 2023 Aug 16;14:1209063. doi: 10.3389/fphar.2023.1209063. eCollection 2023. PMID 37663252
- [Background] Povoa FCC, Cardinal-Fernandez P, Maia IS, Reboredo MM, Pinheiro BV. Effect of antibiotics administered via the respiratory tract in the prevention of ventilator-associated pneumonia: A systematic review and meta-analysis. J Crit Care. 2018 Feb;43:240-245. doi: 10.1016/j.jcrc.2017.09.019. Epub 2017 Sep 18. PMID 28942198
- [Background] Lu Q, Luo R, Bodin L, Yang J, Zahr N, Aubry A, Golmard JL, Rouby JJ; Nebulized Antibiotics Study Group. Efficacy of high-dose nebulized colistin in ventilator-associated pneumonia caused by multidrug-resistant Pseudomonas aeruginosa and Acinetobacter baumannii. Anesthesiology. 2012 Dec;117(6):1335-47. doi: 10.1097/ALN.0b013e31827515de. PMID 23132092
- [Background] Biswas S, Brunel JM, Dubus JC, Reynaud-Gaubert M, Rolain JM. Colistin: an update on the antibiotic of the 21st century. Expert Rev Anti Infect Ther. 2012 Aug;10(8):917-34. doi: 10.1586/eri.12.78. PMID 23030331
- [Background] Yu Z, Qin W, Lin J, Fang S, Qiu J. Antibacterial mechanisms of polymyxin and bacterial resistance. Biomed Res Int. 2015;2015:679109. doi: 10.1155/2015/679109. Epub 2015 Jan 15. PMID 25664322
- [Background] Zhang X, Cui X, Jiang M, Huang S, Yang M. Nebulized colistin as the adjunctive treatment for ventilator-associated pneumonia: A systematic review and meta-analysis. J Crit Care. 2023 Oct;77:154315. doi: 10.1016/j.jcrc.2023.154315. Epub 2023 Apr 28. PMID 37120926
- [Background] Hu JN, Hu SQ, Li ZL, Bao C, Liu Q, Liu C, Xu SY. Risk factors of multidrug-resistant bacteria infection in patients with ventilator-associated pneumonia: A systematic review and meta-analysis. J Infect Chemother. 2023 Oct;29(10):942-947. doi: 10.1016/j.jiac.2023.06.008. Epub 2023 Jun 13. PMID 37321291
- [Background] Ranzani OT, Niederman MS, Torres A. Ventilator-associated pneumonia. Intensive Care Med. 2022 Sep;48(9):1222-1226. doi: 10.1007/s00134-022-06773-3. Epub 2022 Jun 30. No abstract available. PMID 35771252
- [Background] Xie J, Yang Y, Huang Y, Kang Y, Xu Y, Ma X, Wang X, Liu J, Wu D, Tang Y, Qin B, Guan X, Li J, Yu K, Liu D, Yan J, Qiu H. The Current Epidemiological Landscape of Ventilator-associated Pneumonia in the Intensive Care Unit: A Multicenter Prospective Observational Study in China. Clin Infect Dis. 2018 Nov 13;67(suppl_2):S153-S161. doi: 10.1093/cid/ciy692. PMID 30423055
- [Background] Ding X, Ma X, Gao S, Su L, Shan G, Hu Y, Chen J, Ma D, Zhang F, Zhu W, Sun G, Meng X, Ma L, Zhou X, Liu D, Du B; China National Critical Care Quality Control Center Group. Effect of ICU quality control indicators on VAP incidence rate and mortality: a retrospective study of 1267 hospitals in China. Crit Care. 2022 Dec 29;26(1):405. doi: 10.1186/s13054-022-04285-6. PMID 36581952
- [Background] Ehrmann S, Barbier F, Demiselle J, Quenot JP, Herbrecht JE, Roux D, Lacherade JC, Landais M, Seguin P, Schnell D, Veinstein A, Gouin P, Lasocki S, Lu Q, Beduneau G, Ferrandiere M, Plantefeve G, Dahyot-Fizelier C, Chebib N, Mercier E, Heuze-Vourc'h N, Respaud R, Gregoire N, Garot D, Nay MA, Meziani F, Andreu P, Clere-Jehl R, Zucman N, Azais MA, Saint-Martin M, Gandonniere CS, Benzekri D, Merdji H, Tavernier E; Reva and CRICS-TRIGGERSEP F-CRIN Research Networks. Inhaled Amikacin to Prevent Ventilator-Associated Pneumonia. N Engl J Med. 2023 Nov 30;389(22):2052-2062. doi: 10.1056/NEJMoa2310307. Epub 2023 Oct 25. PMID 37888914
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Metersky ML, Kalil AC. Management of Ventilator-Associated Pneumonia: Guidelines. Infect Dis Clin North Am. 2024 Mar;38(1):87-101. doi: 10.1016/j.idc.2023.12.004. PMID 38280768